CLINICAL TRIAL: NCT07180251
Title: Impact of Glycemic Variability on Diabetes Self-care, Glycated Hemoglobin, Diabetes Distress, Fatigue, and Quality of Life in People With a Dual Diagnosis of Gastrointestinal Cancer and Diabetes After Surgery
Brief Title: Impact of Glycemic Variability on People With Gastrointestinal Cancer and Diabetes After Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202501119RIND
Record Dates: First submitted 2025-09-09; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Melletus; Gastrointestinal Cancers
Keywords: diabetes mellitus; gastrointestinal cancer; glycemic variability
MeSH Terms: conditions — Gastrointestinal Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: In phase 1, a longitudinal, observational design will be used to examine the link between glycemic variability and its predictors and outcomes. In phase 2, a randomized controlled trial design, recruiting participants from three GI surgical OPDs at a medical center in northern Taiwan, will be used. Specifically, after completing the pre-tests, stratification of colorectal, gastric, and pancreatic cancer patients will be performed according to the proportionate of new cases for colorectal, gastric, and pancreatic cancer reported in the National Cancer Registry. investigators will recruit participants who are planning to undergo GI cancer surgery, and participants in the experimental group will begin the 8-week intervention at 3 months postsurgery. Pre-tests will be performed before intervention (T0). The short-term, mid-term, and long-term effects will be measured at 8 weeks (T1; immediately after program completion), 3 months (T2), and 6 months (T3) post-intervention, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care + CARE program (Experimental): For the intervention group, participants will receive usual care and will be scheduled for the first in-person session of the CARE program after completing the T0 questionnaires, and will complete the outcome measurements using structured questionnaires at T1: Post-test 1 (5 months after surgery), T2: Post-test 2(6 months after surgery), and T3: Post-test 3(9 months after surgery).
  Interventions: Behavioral: CARE program; Other: Usual Care
- Usual Care (Other): The control group will receive usual care. After obtaining the participants' written informed consent, baseline data will be collected (T0), and will complete the outcome measurements using structured questionnaires at T1: Post-test 1 (5 months after surgery), T2: Post-test 2 (6 months after surgery), and T3: Post-test 3 (9 months after surgery).
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: CARE program — The CARE program is an 8-week intervention using reflection assisted with CGM. The Abbott factory-calibrated Freestyle Libre Flash Glucose Monitoring (Freestyle Libre 2) system will be used to evaluate glycemic variability.
  Arms: Usual care + CARE program
Other: Usual Care — Usual care means the participants will receive care from their primary care physicians and nurses during clinic visits at the surgical OPD.

SUMMARY:
In study phase 1, the investigators will prospectively examine the factors related to post-operative glycemic variability and its effect on outcomes in people with both DM and GI cancer after surgery. The study will also qualitatively understand the glycemic variability experiences and their associated symptoms and outcomes in people with both DM and GI cancer. In study phase 2, the investigators will develop and test the effects of the CGM-Assisted Reflection Education (CARE) program on adults with both DM and GI cancer post-surgery.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) often coexists with gastrointestinal (GI) cancer, and poor post-operative glycemic control is hypothesized as a major cause of patients' worse health-related outcomes. No study to date has developed and tested a program that focuses on improving DM self-care through glycemic variability reflection using continuous glucose monitoring (CGM) in people with both GI cancer and DM after surgery. This study aims to (1) prospectively examine the relationships among factors influencing glycemic variability and outcomes (DM self-care, HbA1c, DM distress, fatigue, and quality of life) in adults with DM and GI cancer during the first year post-surgery; (2) qualitatively explore the glycemic variability experiences; and (3) develop and test the effects of the CGM-Assisted Reflection Education (CARE) program on DM self-care and the secondary outcomes. This study consists of two phases. Phase one will utilize a longitudinal mixed-methods design with 200 participants recruited from GI surgical outpatient departments, collecting data via structured questionnaires at four time points: before surgery, 3, 6, and 12 months post-surgery. Data will be analyzed using SPSS version 28 and Mplus version 8.6 under a structural equation modeling approach. A subsample of 21 participants will undergo semi-structured interviews for qualitative insights. In study phase two, the CARE program will be developed and tested using a randomized controlled trial design. A total sample of 60 participants (30 in each group) will be recruited and randomly assigned in a 1:1 ratio to the experimental and the control group. The experimental group will receive usual care plus the CARE program. The control group will receive usual care. Outcomes will be measured using the same set of questionnaires from phase one, and the data will be collected pre-intervention, 8 weeks, 3-, and 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are planning to undergo GI cancer surgery according to their physician's advice
* Diagnosed with diabetes mellitus
* Aged 18 or above
* Can communicate in Mandarin or Taiwanese
* Agree to participate and sign the informed consent form

Exclusion Criteria:

* People who are under active treatment for cancer other than GI cancer
* Have a cognitive impairment
* Do not know that they have GI cancer
* Have medical-grade adhesives-related allergy (e.g., redness, swelling, heat, pain, itching, blisters or rash)
* Diagnosed with thrombocytopenia or blood coagulation dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-Care of Diabetes Inventory | before surgery (T0), 3 (T1), 6 (T2), and 12 (T3) months post-surgery
  The Self-Care of Diabetes Inventory total score ranges from 40 to 200, and higher scores mean better diabetes self-care.

SECONDARY OUTCOMES:
Diabetes Distress Scale | before surgery (T0), 3 (T1), 6 (T2), and 12 (T3) months post-surgery
  The Diabetes Distress Scale ranges from 15 to 90, with higher scores indicating worse diabetes distress.
Fatigue Symptom Inventory | before surgery (T0), 3 (T1), 6 (T2), and 12 (T3) months post-surgery
  The Fatigue Symptom Inventory total score ranges from 0 to 127, with higher scores indicating worse fatigue.
European Organisation for Research and Treatment of Cancer Quality of Life | before surgery (T0), 3 (T1), 6 (T2), and 12 (T3) months post-surgery
  The global health status/quality of life subscale of the European Organisation for Research and Treatment of Cancer Quality of Life scale ranges from 1 to 7, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Ju Kuo, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No